CLINICAL TRIAL: NCT00140803
Title: A Randomized, Single-Masked, Multi-Center, Phase 2 Evaluation Of The Effect Of PDT Using Visudyne In Combination With Intravitreal Injection Of Either 0 mg, 1mg or 4mg of Kenalog In Subfoveal Occult & Minimally Classic CNV Secondary To ARMD
Brief Title: Study Of Combined VISUDYNE Therapy With Kenalog In CNV Secondary To Age-Related Macular Degeneration
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Manhattan Eye, Ear & Throat Hospital (Other)
Collaborators: Novartis (Industry); QLT Inc. (Industry)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: VISTA
Expanded Access: Available
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2007-07-12 (Estimated); Status verified 2007-07

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Verteporfin; Triamcinolone Acetonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Visudyne
Drug: Kenalog

SUMMARY:
To determine whether VISUDYNE therapy in combination with 4 mg intravitreal triamcinolone will reduce the average loss from baseline of best corrected visual acuity (BCVA) as compared with Visudyne therapy without intravitreal triamcinolone at 12 months in subjects with occult subfoveal and minimally classic subfoveal CNV secondary to AMD. The intravitreal triamcinolone will be given as either a 1 mg or 4 mg dose. This study will also evaluate the safety of Visudyne therapy in combination with intravitreal triamcinolone. An interim statistical readout will be performed when the first 60 patients have completed 6 months of follow-up evaluation.

DETAILED DESCRIPTION:
This is a randomized, single-masked (VA examiners, angiographic graders), multi-center, Phase 2 study with 3 arms comparing VISUDYNE therapy in combination with intravitreal injection of either a 1 mg or 4 mg of triamcinolone with VISUDYNE therapy without intravitreal triamcinolone in a 1:1:1 ratio.

Re-treatment may be administered at 3 month intervals ( 14 days) if evidence of CNV leakage is detected by fluorescein angiography.

At baseline and at 3 month (+ 14 days) intervals patients will undergo the following assessments: ophthalmic examination, best corrected visual acuity, fluorescein angiography, and color fundus photography. The eligibility criteria for inclusion into the study and re-treatment of patients will be based on fluorescein angiography. Patients receiving treatment at day-1, week-3, and week-6 following the treatment will have best corrected ETDRS visual acuity testing and ophthalmic. Those patients not being re-treated will have will have best corrected ETDRS visual acuity testing and ophthalmic examination at week-6 following the re-treatment evaluation visit.

Adverse events will be assessed throughout the study.

Expected time for recruitment is 6 months; all patients will be followed for the period of 12 months in the study

ELIGIBILITY:
Inclusion Criteria:

* • Age 50 years or older

  * Subfoveal CNV secondary to age-related macular degeneration
  * Area of the CNV at least 50% of the area of the total neovascular lesion
  * The lesion is either minimally classic or occult with no classic
  * If the lesion is occult with no classic then subjects must have presumed recent disease progression in the study eye in the judgment of the Investigator and as defined by presence of blood associated with the lesion or vision loss or lesion growth reported or objectively recorded within the preceding 3 months before randomization to treatment
  * Baseline BCVA score between 73 and 19 letters on the ETDRS scale (approximately 20/40 to 20/400)
  * Lesion size < 5400 microns
  * Ability and willingness to provide written informed consent.

Exclusion Criteria:

* Subjects may not be randomized to treatment if they:

  1. Have evidence of predominantly classic CNV, clinically significant intraocular inflammation, angioid streaks, presumed ocular histoplasmosis syndrome, axial myopia greater than -6 diopters, or other precursors of choroidal neovascularization
  2. Have additional eye disease that compromises the visual acuity of the study eye.
  3. Are receiving or require chronic concomitant therapy with systemic or topical ocular corticosteroids or NSAIDS. Chronic concomitant therapy is defined as multiple doses taken daily for 3 or more consecutive days at any time during the course of the 12-month study). A low dose (up to 100 mg po qd) of aspirin (ASA) taken for prophylaxis of MI and/or stroke is permitted during the study.
  4. Are using coumadin.
  5. Have known hypersensitivity to verteporfin or triamcinolone
  6. Have CNV that does not involve the geometric center of the foveal avascular zone, as determined by color photography and fluorescein angiography
  7. Are unable to be photographed to document CNV, e.g. due to media opacity, allergy to fluorescein dye or lack of venous access
  8. Have lens opacities which, in the investigator's opinion, would progress during the course of the study and would affect central vision in the study eye. Such cataracts may be removed at least 2 months before entering the subject in the study
  9. Have a history of treatment for CNV, other than confluent laser photocoagulation, in the study eye (e.g., PDT, submacular surgery, radiotherapy or macular scatter "grid" laser photocoagulation
  10. Are participating in another clinical trial requiring follow-up examinations or are receiving or have received any experimental treatment for CNV or any other investigational new drug within 12 weeks prior to the start of study treatment
  11. Have an intraocular pressure greater than 21 mm Hg on or off medication on entry to the study.
  12. Have received prior treatment with another anti-angiogenic compound (e.g., Sandostatin®, LY333531, Macugen, RhuFab, etc.) within 6 months prior to screening
  13. Are unwilling or unable to follow or comply with all study-related procedures.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2003-10; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to determine the effect of Visudyne therapy in combination with 4 mg intravitreal triamcinolone on the mean change in BCVA at Month 12. | 12 months

SECONDARY OUTCOMES:
• Proportion of patients having a 15 letter (3 lines) loss or more in BCVA | 12 months
• Proportion of patients having a 15 letter (3 lines) improvement or more in BCVA | 12 months
• Proportion of patients requiring re-treatment at any time during the study | 12 months
• The number of re-treatments required | 12 months
• Difference in treatment effect between 1 mg and 4 mg of triamcinolone acetonide | 12 months
• The change in MNREAD score | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard F. Spaide, MD, Principal Investigator — Manhattan Eye, Ear & Throat Hospital
Locations (2):
- Manhattan Eye, Ear & Throat Hospital, New York, New York, United States
- Vh/UBC Eye Care Centre, Vancouver, British Columbia, Canada